CLINICAL TRIAL: NCT04664712
Title: Efficacy of Focused Shock Waves Combined With Adjuvant Therapy With Tendon Supplement in the Treatment of Plantar Fasciitis: a Prospective Randomized Study
Brief Title: Efficacy of Focused Shock Waves Combined With Adjuvant Therapy With Tendon Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWT-TP
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Fasciitis, Plantar
Keywords: focused shock waves; tendinitis; natriuretics
MeSH Terms: conditions — Fasciitis, Plantar; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- shock wave (Active Comparator)
  Interventions: Device: Focused shock wave
- shock wave and tendon supplement (Active Comparator)
  Interventions: Dietary Supplement: Tendisulfur Pro; Device: Focused shock wave

INTERVENTIONS:
Dietary Supplement: Tendisulfur Pro — Dietary supplement based on Methylsulfonylmethane (2.5 g), hydrolyzed collagen (1 g), L-arginine (1 g), L-lysine (500 mg), Vitamin C (500 mg), Bromelain (200 mg), Chondroitin sulfate (150 mg), Glucosamine (150 mg) [17, 18], dry extracts of turmeric (100 mg), Boswellia (100 mg) and Myrrh (50 mg)
  Arms: shock wave and tendon supplement
Device: Focused shock wave — We delivered 2000 shots per session using a low/medium energy level (range between 0.01 and 0.175 milliJoule/mm2) depending on the patient's tolerance during treatment with a frequency of 4 Hz.

SUMMARY:
Physical treatment with focused shock waves is effective in the treatment of tendonitis. Food supplements could facilitate the healing of tendinopathies when combined with shock wave therapy.

DETAILED DESCRIPTION:
A single-blind, randomized prospective study (level of evidence IB) was designed. Patients with plantar fasciitis were recruited and randomized to group A and group B. Group A was treated with focused shock waves alone and group B with a combination of focused shock waves and tendon supplement. Pain remission (primary endpoint) and functional recovery (secondary endpoint) are monitored in both groups at three time points (Months 0, 3, and 6).

ELIGIBILITY:
Inclusion Criteria:

* plantar heel pain diagnosed clinically and instrumentally (ultrasound) as plantar fasciitis, that has not responded to conservative treatment for at least six months;

Exclusion Criteria:

* History of previous fractures or ankle and heel surgery;
* Recurrence of previous local painful episodes;
* Lesion of the plantar fascia on US examination;
* Presence of pathologies that affect the function of the foot (lumbar radiculopathy, Achilles tendinitis, Morton's neuroma, etc.);
* Chronic inflammatory conditions such as psoriasis, psoriatic arthritis, spondyloarthritis, ankylosing spondylitis, rheumatoid arthritis, chronic inflammatory bowel disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Score (VAS) | T0 (recruitment); T1 (three months)
  The pain was quantified using the VAS scale with the scores ranging between 0 (no pain) and 10 (worst imaginable pain).
Change in Visual Analogue Score (VAS) | T1 (three months); T2 (six months)
  The pain was quantified using the VAS scale with the scores ranging between 0 (no pain)

SECONDARY OUTCOMES:
Change in American Foot & Ankle Score (AOFAS) | T0 (recruitment); T2 (six months)
  The scores ranging between 100 (no disability) and 0 (maximum disability)
Change in Foot Function Index (FFI) | T0 (recruitment); T2 (six months)
  The scores ranging between 100 (no disability) and 0 (maximum disability).
Roles & Maudsley (R&M) | T1 (three months)
  Monitorization of the patient's perception of improvement, with the scores ranging from 1 (excellent) to 4 (minimum).
Roles & Maudsley (R&M) | T2 (six months)
  Monitorization of the patient's perception of improvement, with the scores ranging from 1 (excellent) to 4 (minimum).

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Moretti, Prof, Principal Investigator — University of Bari Aldo Moro
Locations (1):
- AOUC Policlinico di Bari - UOC Ortopedia e Traumatologia, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
No sharing